CLINICAL TRIAL: NCT03368326
Title: Use of Critical-Care Pain Observation Tool and Bispectral Index for Detection of Pain in Brain Injured Patients：A Prospective Observational Study
Brief Title: Use of Critical-Care Pain Observation Tool and Bispectral Index for Detection of Pain in Brain Injured Patients
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Director of Intensive Care Unit, Capital Medical University
Other Study IDs: CHDR-2014-2-2041
Record Dates: First submitted 2017-12-04; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Intensive Care; Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Critical-Care Pain Observation Tool (CPOT) — The CPOT includes 4 behaviors: (1) facial expression, (2) body movements, (3) compliance with the ventilator, and (4) muscle tension. Each behavior is rated from 0 to 2 for a possible total score ranging from 0 to 8.
  Other Names: Bispectral Index (BIS)

SUMMARY:
Brain injured patients are at high risk of pain due to the illness itself and a variety of nociceptive procedures in intensive care unit. Since the disorder of consciousness, speech, and movement, it is usually difficult for them to self-report the presence of pain reliably. The Critical-Care Pain observation Tool (CPOT) has been recommended for clinical use in the critically ill patients when self-report pain is unavailable. Besides, it seems that the bispectral index (BIS), a quantified electroencephalogram instrument, can be used for pain assessment along with the CPOT tool in some nonverbal critical ill patients (e.g., intubated and deep sedation). However, the validity and reliability of CPOT and BIS for pain assessment in brain injured patients are still uncertain so far. So the aim of this research is to investigate the value of CPOT and BIS for pain evaluation in this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

* patients with brain injury and artificial airway

Exclusion Criteria:

* age under 18 years,
* quadriplegia,
* administration of paralytic medications within 24 hours,
* if the patient failed the quality test of BIS signal,
* impending death,
* be included in any other research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with brain injury and artificial airway
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Changes of the Critical-Care Pain Observation Tool (CPOT) scores | 1.Before nociceptive/non-nociceptive procedure; 2.Within the first 5 minutes after nociceptive/non-nociceptive procedure.
  The CPOT includes 4 behaviors: (1) facial expression, (2) body movements, (3) compliance with the ventilator, and (4) muscle tension. Each behavior is rated from 0 to 2 for a possible total score ranging from 0 to 8.
Changes of the bispectral Index (BIS) value | 1.Before nociceptive/non-nociceptive procedure; 2.Within the first 5 minutes after nociceptive/non-nociceptive procedure.
  The BIS monitor is a noninvasive technology, which measures different electrocortical indices through electrodes placed on the patient's forehead. Its main variable, the BIS index, consists of a single number computed from a complex algorithmic equation based on the EEG data. Its value can range from 0 (complete EEG suppression) to 100 (fully awake).

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Intensive care unit, Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- Intensive care unit, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided